CLINICAL TRIAL: NCT04048369
Title: Impact Study of a Rapid Diagnosis of Influenza in the Emergency Medical Service During the 2018-2019 Epidemic Season
Brief Title: Impact of Influenza/RSV PCR Point-of-care Testing in the Emergency Medical Service.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: RBHP 2018 HENQUELL; 2018-A02478-47 (Other: ANSM)
Record Dates: First submitted 2019-07-26; First posted 2019-08-07 (Actual); Last update posted 2019-08-07 (Actual); Status verified 2019-06

CONDITIONS: Influenza
Keywords: influenza; point-of-care testing; polymerase chain reaction; emergency medicine
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Point-of-care testing arm (Experimental): for patients randomized to the Point-of-care testing arm, nurse will perform influenza and RSV testing using an FDA-approved point-of-care device (Cepheid Xpert® Xpress Flu/RSV) in the ED, 24/24, 7/7.
  Interventions: Diagnostic Test: Rapid diagnosis of influenza in the emergency medical service
- Core Lab testing arm (Active Comparator): for patients randomized to the Core lab testing arm, influenza/RSV PCR will be performed in the core virology laboratory using Simplexa Flu A/B and RSV direct (r) assay (Diasorin), during working hours (8 am-6pm Monday to Friday, 8 am-5pm the Saturday)
  Interventions: Diagnostic Test: Rapid diagnosis of influenza in the emergency medical service

INTERVENTIONS:
Diagnostic Test: Rapid diagnosis of influenza in the emergency medical service — Comparison at the University Hospital of Clermont-Ferrand of a test performed in the Adult Emergencies Department by the nursing staff (point-of-care testing) to a test carried out in the core laboratory (classical testing).

SUMMARY:
The purpose of the study is to compare Emergency Department patients who undergo influenza and RSV PCR testing using an FDA-approved point-of-care device (Cepheid Xpert® Xpress Flu/RSV) located in the ED, to patients who undergo influenza and RSV PCR testing at the core laboratory.

The principal purpose is to determine if the time spent in the ED is different in the group undergoing POC influenza testing compared to those undergoing laboratory-based influenza testing.

DETAILED DESCRIPTION:
* This study will be conducted during the influenza's epidemic season. The start and the end of this study will be determined using national epidemic bases (national reference center for inluenza in Lyon).
* Collection of consent of eligible patients after medical information by a senior emergency physician
* Sampling = nasopharyngeal swabbing for all patients using usual testing or point-of-care testing
* first arm : performing the test at the adult emergency department 24h/24
* second arm : sending the test to the virology laboratory and realization during working hours
* Collection of clinical data : a specific standardized questionnaire is used, as soon as the patient is included and until he leaves the emergency medical service, to collect clinical data and the time taken to take care of the patient

In order to reduce the bias of this study, it has been established :

After verification of the eligibility criteria and obtaining the written consent of the patient, a randomization procedure will be initiated for the patient. Randomization will be centralized at the DRCI of Clermont-Ferrand University Hospital. Patients will be randomly assigned to one of the study groups by means of individual block randomization. A document describing the randomization procedure will be kept confidentially in the DRCI of Clermont-Ferrand University Hospital;

- The collection of data will be prospective.

A listing of patients opposing to the study's participation to verify that their characteristics are homogeneous to the general population The choice of the Genexpert® automaton used in the "point of care testing" arm whose principle of operation requires a minimum of manipulations (<2 minutes) and does not generate inter-operator variability Statistical analyzes will be performed with the Stata software (version 13, StataCorp, College Station). All statistical tests will be carried out at the risk of error of the first species α of 5%. Part of the analysis of the secondary endpoints should be primarily exploratory in nature. As discussed by Feise in 2002 (Feise RJ, Do 2: 8), the adjustment of the risk of error of 1st species will not be proposed systematically, but case by case in view of clinical considerations and not just statistical ones.

Continuous variables will be presented as mean and standard deviation, subject to the normality of their distribution (Shapiro-Wilk test if necessary). In case of non-normality, they will be presented as median, quartiles, and extreme values. The qualitative variables will be expressed in numbers and percentages associated. Graphic representations will be associated with these analyzes as much as possible.

ELIGIBILITY:
Inclusion criteria :

* 18 years old and older
* coming in the emergency medical service
* during the influenza epidemic period
* with influenza symptoms
* whose support requires virologic confirmation
* people having given their consent

Exclusion criteria :

* pregnant or breast feeding women
* patient unable to give consent
* tutorship or curatorship or under the protection of justice
* patient non registered in the social security system

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 431 (Actual)
Dates: Start 2019-01-17 (Actual); Primary Completion 2019-03-14 (Actual); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Time of care in the adult emergency department | through study completion, an average of 1 week
  Emergency care time, calculated from the time of first medical-care contact to the time of release of the adults emergency department.
  This time will be calculated from the data collected on the standardized questionnaire

SECONDARY OUTCOMES:
Prescription of antibiotics initiated at the adults emergency department | within 72 hours after taking care of the patient
  nature of antibiotics
Duration of the prescription of antibiotics initiated at the adults emergency department | within 72 hours after taking care of the patient
  duration of treatment (day)
Posology of antibiotics initiated at the adults emergency department | within 72 hours after taking care of the patient
  posology (mg)
Costs of antibiotics initiated at the adults emergency department | within 72 hours after taking care of the patient
  associated costs (euros)
Prescription of antiviral initiated in adults emergency department | within 72 hours after taking care of the patient
  nature of antiviral prescription
Duration of the specific antiviral prescription initiated in adults emergency department | within 72 hours after taking care of the patient
  duration of treatment (day)
Costs of specific antiviral prescription initiated in adults emergency department | within 72 hours after taking care of the patient
  associated costs (euros)
Type of prescription of imaging tests at the adults emergency department | within 72 hours after taking care of the patient
  type of examinations related to the patient respiratory pathology
Number of prescription of imaging tests at the adults emergency department | within 72 hours after taking care of the patient
  Number of examinations related to the patient respiratory pathology
Costs of the prescription of imaging tests at the adults emergency department | within 72 hours after taking care of the patient
  Costs of examinations related to the patient respiratory pathology (euros)
Type of prescription of biology examinations | within 72 hours after taking care of the patient
  type of laboratory examinations related to respiratory pathology
Number of prescription of biology examinations | within 72 hours after taking care of the patient
  Number of laboratory examinations related to respiratory pathology
Costs of prescription of biology examinations | within 72 hours after taking care of the patient
  Costs of laboratory examinations related to respiratory pathology (euros)

CONTACTS AND LOCATIONS:
Overall Officials: Cécile Henquell, PU-PH, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU de Clermont-Ferrand, Clermont-Ferrand, Auvergne, France

REFERENCES:
- [Background] Soto M, Sampietro-Colom L, Vilella A, Pantoja E, Asenjo M, Arjona R, Hurtado JC, Trilla A, Alvarez-Martinez MJ, Mira A, Vila J, Marcos MA. Economic Impact of a New Rapid PCR Assay for Detecting Influenza Virus in an Emergency Department and Hospitalized Patients. PLoS One. 2016 Jan 20;11(1):e0146620. doi: 10.1371/journal.pone.0146620. eCollection 2016. PMID 26788921
- [Background] Trabattoni E, Le V, Pilmis B, Pean de Ponfilly G, Caisso C, Couzigou C, Vidal B, Mizrahi A, Ganansia O, Le Monnier A, Lina B, Nguyen Van JC. Implementation of Alere i Influenza A & B point of care test for the diagnosis of influenza in an ED. Am J Emerg Med. 2018 Jun;36(6):916-921. doi: 10.1016/j.ajem.2017.10.046. Epub 2017 Oct 18. PMID 29137903
- [Background] Brendish NJ, Malachira AK, Armstrong L, Houghton R, Aitken S, Nyimbili E, Ewings S, Lillie PJ, Clark TW. Routine molecular point-of-care testing for respiratory viruses in adults presenting to hospital with acute respiratory illness (ResPOC): a pragmatic, open-label, randomised controlled trial. Lancet Respir Med. 2017 May;5(5):401-411. doi: 10.1016/S2213-2600(17)30120-0. Epub 2017 Apr 6. PMID 28392237
- [Background] Ho YII, Wong AH, Lai RWM. Comparison of the Cepheid Xpert Xpress Flu/RSV Assay to in-house Flu/RSV triplex real-time RT-PCR for rapid molecular detection of Influenza A, Influenza B and Respiratory Syncytial Virus in respiratory specimens. J Med Microbiol. 2018 Nov;67(11):1576-1580. doi: 10.1099/jmm.0.000841. Epub 2018 Sep 12. PMID 30207514
- [Background] Banerjee D, Kanwar N, Hassan F, Essmyer C, Selvarangan R. Comparison of Six Sample-to-Answer Influenza A/B and Respiratory Syncytial Virus Nucleic Acid Amplification Assays Using Respiratory Specimens from Children. J Clin Microbiol. 2018 Oct 25;56(11):e00930-18. doi: 10.1128/JCM.00930-18. Print 2018 Nov. PMID 30185508
- [Background] Bennett S, MacLean A, Gunson R. Verification of Cepheid Xpert Xpress Flu/RSV assay for use with gargle samples, sputa and endotracheal secretions. J Hosp Infect. 2019 Jan;101(1):114-115. doi: 10.1016/j.jhin.2018.07.016. Epub 2018 Jul 17. No abstract available. PMID 30026005
- [Background] Popowitch EB, Miller MB. Comparison of the Xpert Flu/RSV XC and Xpress Flu/RSV Assays. J Clin Microbiol. 2018 Jul 26;56(8):e00278-18. doi: 10.1128/JCM.00278-18. Print 2018 Aug. PMID 29769281
- See also: Procédure actualisée de prise en charge globale d'un patient suspect de grippe saisonnière — http://www.infectiologie.com/UserFiles/File/medias/coreb/grippe/proced-grippe-saison-coreb-site-15fev16-1.pdf